CLINICAL TRIAL: NCT02927678
Title: Assessment of White Blood Cell SPECT/CT in Monitoring Antibiotic Treatment in Patients With Diabetic Foot Osteomyelitis
Brief Title: White Blood Cell SPECT/CT and Diabetic Foot Osteomyelitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0597
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-09

CONDITIONS: Diabetic Foot Osteomyelitis
Keywords: Diabetic foot; Osteomyelitis; Antibiotic treatment; White Blood Cell SPECT/CT
MeSH Terms: conditions — Diabetic Foot; Osteomyelitis | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetic patients with osteomyelitis: Patients with a clinical and radiological diagnosis of osteomyelitis were included in two diabetic centers
  Interventions: Other: white blood cell SPECT/CT (Single Photon Emission Computed Tomography/Computed Tomography) imaging

INTERVENTIONS:
Other: white blood cell SPECT/CT (Single Photon Emission Computed Tomography/Computed Tomography) imaging

SUMMARY:
Osteomyelitis is a risk factor for lower extremity amputation in diabetic people. Antibiotic therapy allows a remission in 60 to 80% of cases. However the optimal duration of antibiotic therapy remains controversy due to the absence of validated marker of osteomyelitis remission. We have previously shown that the negativity of white blood cell SPECT/CT (Single Photon Emission Computed Tomography/Computed Tomography) imaging at the end of treatment allowed to predict remission of osteomyelitis at 1 year in all cases. A positive imaging was associated with recurrence in 70% of cases. The aim of our study was to evaluate prospectively the interest of white blood cell SPECT/CT to set the duration of antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Diabetes
* Osteomyelitis defined by soft tissue infection and/or positive probe-to-bone test and suggestive signs of osteomyelitis on plain-X-Ray

Exclusion Criteria:

- Indication for acute surgical bone resection or amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a clinical and radiological diagnosis of osteomyelitis were included in two diabetic centers
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Rate of remission of osteomyelitis at one year after the cessation of antibiotic treatment, evaluated by white blood cell SPECT/CT (Single Photon Emission Computed Tomography/Computed Tomography). | one year after the end of the antibiotic treatment
  The outcome measure was reviewed by patient examination at least 12 months after completion of antibiotic treatment. A remission was defined by :
  * the absence of recurrent infection at the initial site
  * no need for surgical bone resection or amputation

SECONDARY OUTCOMES:
Rate of osteomyelitis remission at one year after a 6 weeks antibiotics duration, evaluated by white blood cell SPECT/CT | one year after the end of the antibiotic treatment
  The outcome measure was reviewed by patient examination at least 12 months after completion of antibiotic treatment. A remission was defined by :
  * the absence of recurrent infection at the initial site
  * no need for surgical bone resection or amputation
Sensibility ration of White Blood Cell SPECT/CT performed at the end of antibiotic treatment to predict the remission of osteomyelitis at one year. | one year after the end of the antibiotic treatment
  Sensibility ratio= number of true positive /number of (true positive+false negative)
Specificity ratio of White Blood Cell SPECT/CT performed at the end of antibiotic treatment to predict the remission of osteomyelitis at one year. | one year after the end of the antibiotic treatment
  Specificity ratio= number of true negative /number of (true negative+false positive)
Positive predictive value of White Blood Cell SPECT/CT performed at the end of antibiotic treatment to predict the remission of osteomyelitis at one year. | one year after the end of the antibiotic treatment
  Positive predictive value = number of true positive / number of (true positive+false positive)
Negative predictive value of White Blood Cell SPECT/CT performed at the end of antibiotic treatment to predict the remission of osteomyelitis at one year. | one year after the end of the antibiotic treatment
  Negative predictive value = number of true negative / number of (true negative+false negative)

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Endocrinologie-Diabétologie-Maladies de la nutrition, GH Sud, Hospices Civils de Lyon, Pierre-Bénite, France

REFERENCES:
- [Derived] Vouillarmet J, Tordo J, Moret M, Michon P, Morelec I. 99mTc-white blood cell SPECT/CT to assess diabetic foot osteomyelitis remission: contribution of semi-quantitative scoring system. Nucl Med Commun. 2021 Jul 1;42(7):713-718. doi: 10.1097/MNM.0000000000001390. PMID 33660690
- [Derived] Vouillarmet J, Moret M, Morelec I, Michon P, Dubreuil J. Application of white blood cell SPECT/CT to predict remission after a 6 or 12 week course of antibiotic treatment for diabetic foot osteomyelitis. Diabetologia. 2017 Dec;60(12):2486-2494. doi: 10.1007/s00125-017-4417-x. Epub 2017 Sep 2. PMID 28866726